CLINICAL TRIAL: NCT00897624
Title: Evaluation of the Detection of Tumor Cells in Bone Marrow and Blood in Patients With Choroid Melanoma
Brief Title: Bone Marrow and Blood Samples From Patients With Metastatic Choroid Melanoma
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000633500; CLCC-IC-Micrometa-Melanome; CLCC-IC-2007-03; INCA-RECF0631
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Intraocular Melanoma
Keywords: metastatic intraocular melanoma; ciliary body and choroid melanoma, medium/large size; ciliary body and choroid melanoma, small size
MeSH Terms: conditions — Uveal Melanoma | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow and blood from patients with cancer may help doctors find out the extent of disease.

PURPOSE: This research study is collecting bone marrow and blood samples from patients with metastatic choroid melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Develop and validate a method of detecting tumor cells in the bone marrow and blood in patients with metastatic choroid melanoma.

OUTLINE: While patients are under general anesthesia for standard treatment of their disease, samples of bone marrow from the iliac crest and blood are collected. Samples are analyzed for the expression of tyrosinase and Melan-a via RT-PCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Choroid melanoma

  * Metastatic disease
* Planning to undergo general anesthesia

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* No contraindications to the collection of a bone marrow sample
* No patient deprived of liberty or under trusteeship (including guardianship)
* No social or psychological situations that preclude the ability to give consent

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Detection of micro-metastatic cells in 20 x 10^6 nucleated cells

CONTACTS AND LOCATIONS:
Overall Officials: Pierre T. Dorval, MD, Principal Investigator — Institut Curie